CLINICAL TRIAL: NCT06822218
Title: High Tone Power Therapy Versus Transcutanuoselectrical Nerve Stimulation on Polyneuropathic Pain in Diabetic Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Zeinab Mahmoud Awad Allah, senior of physiotherapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T/REC/012/003905
Record Dates: First submitted 2022-11-23; First posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Diabete Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- High tone power therapy (Experimental): 30 type 2 diabetic patients with diabetic polyneuropathy. Theses patients will receive High tone power therapy
  Interventions: Device: high tone power therapy
- TENS (Active Comparator): 30 type 2 diabetic patients with diabetic neuropathy. These patients will receive TENS
  Interventions: Device: TENS

INTERVENTIONS:
Device: high tone power therapy — patients will be assigned into 2 groups with pre and post treatment protocol application. all patients will be thoroughly evaluated before and after treatment protocol application.
  Arms: High tone power therapy
Device: TENS — These patients will receive TENS with applied frequencies range from 2 to 120 Hz. for 3 times per week for 30 minutes every session during 3 months of intervention in addition to medications.
  Arms: TENS

SUMMARY:
the results of this study may provide an easy non pharmacological modality for dealing with diabetic polyneuropathic pain. Also, the outcome of this study will guide physiotherapists to develop a new noninvasive treatment modality that may improve patient symptoms and promotes their social participation , this in turn may add to clinical role played by therapists in management of diabetic polyneuropathy. In Addition, increased knowledge of the influence of High tone power therapy on neuropathic pain

DETAILED DESCRIPTION:
This study will be carried out on sixty diabetic male patients with polyneuropathy with ages 50-60 years . Patient will be randomly assigned to two grouos. group A will include 30 type 2 diabetic patients with diabetic polyneuropathy. Theses patients will receive High tone power therapy with Frequencies continuously will be scanned from 4096 Hz to 31768 Hz, allowing for a much higher power of up to 5000 mW to be introduced for 3 times per week, for 3 months for 30 minutes every session.

Group B :

This group will include 30 type 2 diabetic patients with diabetic neuropathy. These patients will receive TENS with applied frequencies range from 2 to 120 Hz. for 3 times per week for 30 minutes every session during 3 months of intervention.

ELIGIBILITY:
Inclusion Criteria:

* The patient selection will be according to the following criteria:

  1. Sixty male patients are diagnosed with diabetic polyneuropathy their ages will be ranged from 50-60 years old.
  2. All patients are ambulant independently.
  3. All patients are under full medical control
  4. HbA1c is ranged from 6.5 : 7 %.
  5. Patients has diabetes more than 10 years.

Exclusion Criteria:

* The participants will be excluded if they meet one of the following criteria:

  1. Psychiatric disorders or seizures.
  2. Visual and auditory impairment or tremors influencing balance.
  3. Other neuromuscular disorders.
  4. Foot deformities and ulcers.
  5. Lower limb operations.
  6. Feverish systemic infection
  7. cardiac pacemaker.

Ages: 50 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Neuropathic pain by DN4 (Douleur Neuropathique en 4 Questions) Questions) | up to 12 weeks
  t is a questionnaire has been developed to facilitate detection of neuropathic pain.total score is 10 .diagnosis of neuropathic pain is 4/10.
Pain pressure threshold algometer | up to 12 weeks
  devices that can be used to identify the pressure and/or force eliciting a pressure-pain threshold. It has been noted in pressure

SECONDARY OUTCOMES:
Glyclated Haemoglobin Level (HbA1c) | up to 12 weeks
  Increasing HbA1c level is significantly associated with increased prevalence of DPN as well as PDPN and non-painful DPN
life disability | up to 12 weeks
  the World Health Organization Quality of Life Brief Version (WHOQOL-BREF) is an abbreviated, 26-item version of the 100-item WHOQOL-100 quality of life measure. The WHOQOL-BREF addresses four quality of life domains: physical health, psychological health, social relationships and environment. Then calculate a domain score for each of the health domains by calculating the average answer points for each domain (sum of answer points divided by number of questions) and multiplying the result by the number 4.

CONTACTS AND LOCATIONS:
Locations (1):
- Om Elmasryeen Genral Hospital, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No